CLINICAL TRIAL: NCT05559164
Title: STACIE: Statins for Reduction of Cardiac Toxicity in Patients Receiving HER2 Targeted Therapy
Brief Title: Statins for Reduction of Cardiac Toxicity in Patients Receiving HER2 Targeted
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Mridula George, MD, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042201; Pro2022000290 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Toxicity; Early-stage Breast Cancer
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Intervention Model Description: Stage I-III HER2positive breast cancer receiving anti-HER2 therapy. Participants will receive Lipitor 40 mg PO daily.
  Anti-HER2 targeted therapy + Lipitor 40mg daily
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anti-HER2 targeted therapy + Lipitor 40mg daily (Experimental): Participants will receive Lipitor 40 mg PO daily while receiving anti-HER2 therapy.
  Interventions: Drug: Lipitor 40mg Tablet

INTERVENTIONS:
Drug: Lipitor 40mg Tablet — LIPITOR® (atorvastatin calcium) tablets will be administered orally as a single dose of 40 mg once daily, with or without food
  Other Names: Atorvastatin Calcium

SUMMARY:
This study proposes that the addition of statins reduces the treatment delays or early discontinuations secondary to cardiotoxicity in patients with Stage I-III HER2 positive breast being treated with anti-HER2 therapy.

DETAILED DESCRIPTION:
A single arm open-label phase 2 study to evaluate the cardioprotective effects of statins in patients with Stage I-III HER2 positive breast cancer receiving HER2 targeted therapy. This study will evaluate the hypothesis that addition of statins will reduce treatment delays/discontinuations related to symptomatic/asymptomatic cardiac dysfunction in patients being treated with anti-HER2 therapy. The long-term goal of this study is to improve disease related outcomes and quality of life measures in patients being treated with anti-HER2 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed diagnosis of Stage I-III female breast cancer (including inflammatory breast cancer)
* Scheduled to receive neoadjuvant/adjuvant HER2 targeted therapy
* Between ≥18 years of age
* Female patients of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment. Female patients must agree to use effective barrier contraception during the period of therapy
* Baseline LVEF ≥ 50%
* Prior cancers allowed if no evidence of disease in last 5 years
* ECOG 0-2
* No prior history of treatment with HER2 targeted therapy or anthracyclines based chemotherapy
* Adequate bone marrow function:

I. ANC ≥ 1000/uL II. platelet count ≥ 100,000/uL III. hemoglobin ≥ 9.0 g/dL

• Adequate hepatic function: I. Total bilirubin ≤ 1.5 X ULN II. AST (SGOT) ≤ 5 X ULN III. ALT (SGPT) ≤ 5 X ULN

* Adequate renal function, Creatinine < 1.5x institutional ULN or calculated creatinine clearance ≥ 50 mL/min as estimated using the Cockcroft-Gault formula
* Ability to understand the nature of this study protocol and give written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Participants with stage IV breast cancer
* Participants currently taking statins
* Uncontrolled hypertension (systolic blood pressure >190 mm Hg or diastolic blood pressure >100 mm Hg)
* No active liver disease
* Current use of CYP 3A4 inhibitors
* Any condition including the presence of laboratory abnormalities, which, in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study
* Life expectancy < 12 weeks
* Pregnancy (positive pregnancy test) or lactation
* Pre-existing sensory neuropathy > grade one
* Has significant cardiovascular disease, such as:

LVEF < 50% at baseline as assessed by ECHO (preferred) i) Class III or Class IV myocardial disease as described by the New York Heart Association ii) Recent history (within 6 months prior to enrollment) of myocardial infarction; or iii) Symptomatic arrhythmia at the time of randomization

* Major surgery without complete recovery in the past four weeks prior to screening
* Concurrent active infection
* Participant with uncontrolled and/ or active infection with HIV, Hepatitis B or Hepatitis C
* Participant who has a history of allergy or hypersensitivity to any of the study drugs
* Participant with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, interstitial pulmonary fibrosis, pulmonary hypersensitivity pneumonitis
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — • Female patients of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment. Female patients must agree to use effective barrier contraception during the period of therapy.
Enrollment: 60 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With at Least One Adverse Event will be measured using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 for five years | Five years
  Adverse events (AEs) will be measured using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 for five years

SECONDARY OUTCOMES:
Patient reported outcome (PRO) for pain measured by the quality of Life questionnaire using PROMIS to measure pain | Baseline, six, twelve and fifteen months
  Quality of Life questionnaire using PROMIS will be administered at baseline, six, twelve and fifteen months

OTHER OUTCOMES:
Patient reported outcome (PRO) for pain measured by the quality of Life questionnaire using PROMIS to measure fatigue | Baseline, six, twelve and fifteen months
  Quality of Life questionnaire using PROMIS will be administered at baseline six, twelve and fifteen months
Patient reported outcome (PRO) for pain measured by the quality of Life questionnaire using PROMIS to measure physical functioning | Baseline, six, twelve and fifteen months
  Quality of Life questionnaire using PROMIS will be administered at baseline six, twelve and fifteen months to measure physical functioning
Patient reported outcome (PRO) for pain measured by the quality of Life questionnaire using PROMIS to measure emotional distress | Baseline, six, twelve and fifteen months
  Quality of Life questionnaire using PROMIS will be administered at baseline six, twelve and fifteen months to measure emotional distress
Patient reported outcome (PRO) for pain measured by the quality of Life questionnaire using PROMIS to measure social participation | Baseline, six, twelve and fifteen months
  Quality of Life questionnaire using PROMIS will be administered at baseline six, twelve and fifteen months to measure social participation

CONTACTS AND LOCATIONS:
Overall Officials: Mridula George, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (10):
- United States (10):
  - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, Hamilton, New Jersey
  - RWJBarnabas Health - - Jersey City Medical Medical, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center, Long Branch, New Jersey
  - Monmouth Community Medical, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: No